**Cover Page** 

Title: A Prospective Study of Evaluation of Operative Duration as a Predictor of Mortality in

Pediatric Emergency Surgery: Concept of 100 Minutes Laparotomy in Resource-limited

Setting

NCT Identifier Number: Not assigned

**Document Date:** 31/03/2017

## **Statistical Analysis Protocol**

Data recording and follow-up progress was done with *SURGILOG*® android application. At the end of the study, the data was analyzed comprehensively and statistical calculations were made. Data analysis was done with *IBM SPSS Statistics*® software version 24. Mean and standard deviation were observed for continuous forms of data like age, operative duration, and so on. Tests of normality in the form of Kolmogorov-Smirnov and Shapiro-Wilk analysis was done. Such data was further evaluated for significance by Wilcoxon-Mann-Whitney U test as the data was found to be having non-Gaussian distribution. Further, binary logistic regression analysis was performed on the data to check for independent associations. A p-value of less than 0.05 was considered statistically significant for all practical applications.